CLINICAL TRIAL: NCT03202576
Title: Nasogastric Tube Securement: Comparison of Standard Practice Versus Nasal Bridle for Pediatric Hospitalized Patients
Brief Title: Nasogastric Tube Securement Comparison Study
Acronym: NTSNB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-0691
Record Dates: First submitted 2017-06-12; First posted 2017-06-28 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Failure to Thrive; Nutritional Deficiency; Constipation; Bowel Obstruction; Feeding and Eating Disorders
Keywords: nasogastric tube; microbridle
MeSH Terms: conditions — Failure to Thrive; Malnutrition; Constipation; Intestinal Obstruction; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Evaluate the securement of the Nasogastric tube either by standard securement or using a Nasal Bridal securement method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasogastric tube standard securement (No Intervention): Standard securement of nasogastric tube with adhesive tape
- Nasogastric Tube Nasal Bridle Securement (Experimental): Securement of NG with AMT Micro Bridle
  Interventions: Device: Nasal Bridle

INTERVENTIONS:
Device: Nasal Bridle — Nasal bridle placement and securement of the tube. Instead of taping the tube to the patient's face, nose or upper lip the bridle is a device whereby a magnetic retrieval system is attached to 1/8 inch umbilical tape which is inserted via the nares, looping around the nasal septum and vomer bone and ending with both ends of the bridle (umbilical tape) secured together and to the feeding tube just outside the nose.
  Other Names: Microbridle
  Arms: Nasogastric Tube Nasal Bridle Securement

SUMMARY:
This study evaluates the use of tape to secure nasogastric tubes compared to securement with a nasal bridle device.

DETAILED DESCRIPTION:
Patients who need to have a tube placed through their nose and into their stomach for medical treatments will sometimes have it accidentally removed. A nasal bridle is a device where a magnetic is used to attach a small piece of cloth tape that loops around the nasal septum bone and secures to the nasal gastric tube to prevent it from being pulled out accidentally.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to Children's Hospital Colorado to:

   * 6th floor surgical inpatient unit, or
   * 8th floor medical inpatient unit, or
   * Heart Institute (Cardiac Intensive Care Unit or Cardiac Progressive Care Unit), or
   * Interventional Radiology.
2. Require a nasogastric or transpyloric tube (Corpak tube or clear feeding tube) for feeding or bowel cleanout.
3. Predicted length of use is at least 48 hours.
4. Newborn up to 21 years of age
5. Have a completed consent for enrollment into the study.

Exclusion Criteria:

1. Burn patients because standard for placement is the nasal bridle;
2. Patients with contraindications for bridle placement , such as

   * mechanical obstruction of the nasal airway
   * facial or nasal fractures
   * fracture of the anterior part of the cranium, or basilar skull fractures
3. Any tubes placed for decompression (i.e. Salem Sump tubes)
4. Nasally intubated, or
5. With CPAP/BiPAP.

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Tube dislodgment | Up to 4 weeks
  Compare the rate/percent of nasogastric tube dislodgement utilizing standard tube securement practice vs. nasal bridle (micro bridle) tube securement device in pediatric hospitalized patients.

SECONDARY OUTCOMES:
Device usability | Up to 4 weeks
  Ease of use of the nasal bridle device
Radiation exposure | Up to 4 weeks
  Number of X-rays to confirm tube placement.
Cost | Up to 4 weeks
  Average costs among groups related to naso-gastric (NG) tube placement and replacement
Restraint use | Up to 4 weeks
  Use of restraints for the purpose of tube protection.
Skin integrity | Up to 4 weeks
  Skin integrity: complications/issues
Patient/Caregiver Satisfaction | Up to 4 weeks
  Patient/caregiver satisfaction with bridle.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Banks (Taubert-Dupey), BSN, Principal Investigator — Childrens Hospital Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bechtold ML, Nguyen DL, Palmer LB, Kiraly LN, Martindale RG, McClave SA. Nasal bridles for securing nasoenteric tubes: a meta-analysis. Nutr Clin Pract. 2014 Oct;29(5):667-71. doi: 10.1177/0884533614536737. PMID 25606648
- [Result] Brugnolli A, Ambrosi E, Canzan F, Saiani L; Naso-gastric Tube Group. Securing of naso-gastric tubes in adult patients: a review. Int J Nurs Stud. 2014 Jun;51(6):943-50. doi: 10.1016/j.ijnurstu.2013.12.002. Epub 2013 Dec 25. PMID 24440003
- [Result] Gunn SR, Early BJ, Zenati MS, Ochoa JB. Use of a nasal bridle prevents accidental nasoenteral feeding tube removal. JPEN J Parenter Enteral Nutr. 2009 Jan-Feb;33(1):50-4. doi: 10.1177/0148607108321704. Epub 2008 Sep 30. PMID 18827069
- [Result] Parks J, Klaus S, Staggs V, Pena M. Outcomes of nasal bridling to secure enteral tubes in burn patients. Am J Crit Care. 2013 Mar;22(2):136-42. doi: 10.4037/ajcc2013105. PMID 23455863